CLINICAL TRIAL: NCT05792293
Title: Role of Statin Therapy in Prevention of Anthracycline-Induced Cardiotoxicity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Lotfy Mohamed, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASUMD45/2021
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Doxorubicin Induced Cardiomyopathy
Keywords: Anthracyclines; Doxorubuicn; Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Fifty female patients diagnosed with breast cancer receiving Anthracycline based chemotherapy
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Control Group (Placebo Comparator): Fifty female patients diagnosed with breast cancer receiving Anthracycline based chemotherapy
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — 40 mg oral dose of atorvastatin , lipid lowering drug with other pleotropic effects
  Arms: Study Group
Other: Placebo — Placebo
  Arms: Control Group

SUMMARY:
This study aims at evaluating the role of Atorvastatin in prevention of Anthracycline induced cardiotoxicity

DETAILED DESCRIPTION:
The study participants are female patients with breast cancer receiving Anthracycline based chemotherapy.

They will be divided into 2 groups , the first group will receive 40 mg oral atorvastatin through out the study , while the other group will receive a placebo.

Full echocardiographic study including 3D echocardiography will be done to all patients before starting their chemotherapy and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with histology proven breast cancer with an indication to primary systemic therapy or adjuvant regimens based on anthracyclines

Exclusion Criteria:

* Patients with impaired LV systolic function (EF below 50%)
* Patients with severe valvular heart disease
* Patients previously diagnosed with coronary artery disease
* Patients with baseline elevated liver enzymes
* Patients with prior chemotherapy or radiation therapy
* Pregnant females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients diagnosed with breast cancer
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of cancer therapy related cardiac dysfunction among the two groups | Six months
  cancer therapy related cardiac dysfunction defined as drop in ejection fraction more than 10% and to a value below 53% assessed by 3D echocardiography

SECONDARY OUTCOMES:
Changes in left ventricular ejection fraction assessed by 3D echocardiography among the two groups | Six months
Changes in left ventricular volumes assessed by 3D echocardiography among the two groups | Six months
Changes in left ventricular diastolic function among the two groups | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed L Mohamed, Master, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided